CLINICAL TRIAL: NCT02833636
Title: Prognostic Value of The Age, Creatinine, and Ejection Fraction Score for Non-infarct-related Chronic Total Occlusion Revascularization After Primary Percutaneous Intervention in Acute ST-elevation Myocardial Infarction Patients: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Xibei Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010cto-1
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cto, Acef Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Successful CTO-PCI group: low ACEF score <1.215 (n = 79), intermediate ACEF score from 1.215 to 1.493 (n=70), and high ACEF score≥1.493 (n=72)
  Interventions: Procedure: ACEF score
- Failed/non-attempted CTO-PCI group: low ACEF score<1.215 (n=45), intermediate ACEF score from 1.215 to 1.493 (n=57), and high ACEF score≥1.493 (n=54).
  Interventions: Procedure: ACEF score

INTERVENTIONS:
Procedure: ACEF score

SUMMARY:
The age, creatinine, and ejection fraction (ACEF) score has been used to evaluate the clinical prognostic to patients who underwent PCI. However, it is not known if ACEF score could evaluate the prognostic of recanalization of non-infarct-related coronary arteries (non-IRA) chronic total occlusions (CTO) in patients who successful underwent primary PCI. The objectivity of current study was to assess the prognostic value of ACEF score in acute ST-segment elevation myocardial infarction (STEMI) patients with non-IRA CTO after successful primary PCI.

ELIGIBILITY:
Among the 2952 patients with STEMI successful treatment by PCI, 395 patients (13.4%) had a non-IRA CTO lesion. 18 patients were excluded from current study as they death within 7 days (n=6) or were not to follow-up (n=7). Due to unavailability of ejection fraction or renal function before CTO-PCI, ACEF score could not be calculated in 5 patients. The remaining 377 patients (95.4%) were finally analyzed in the study. 279 patients performed a staged CTO-PCI attempt(ranging 7-28 days) and was successful in 221 of them. Due to low possibility of PCI success or patients refused to perform PCI, 98 patients did not undergo the PCI attempt. The patients were then divided into successful CTO-PCI group (221 patients) and failed/ non-attempted CTO-PCI group (156 patients).

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between January 2006 to December 2013, a total of 2952 consecutive and unselected acute STEMI patients were admitted to our hospital and treated with successful primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 2952 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary end point | 1 year
  Primary end point in the current study was a composite of all-cause death, nonfatal myocardial infarction, ischemia-driven coronary revascularization and hospitalization for heart failure at 1year.